CLINICAL TRIAL: NCT03191747
Title: Examining the Association Between Adherence to Masculine Norms and Skin Care Knowledge, Attitudes, and Behaviors in Adult Men
Brief Title: Masculine Norms and Skin Care Knowledge, Attitudes, and Behaviors
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: STU00205216
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Social Norms
Keywords: Masculine Norms; Skin Care; Gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Examining whether men with greater Avoidance to Femininity subscores using the Male Role Norms Inventory - Short Form will demonstrate differences in skin care knowledge, attitudes, and behaviors, compared to men with lower subscores.

DETAILED DESCRIPTION:
This purpose of this study is to examine whether a man's adherence to traditional masculine norms correlates with his skin care attitudes or behaviors. A stronger understanding of these associations may enable dermatologists to better understand their patient's perception of skin care. The utility of this knowledge lies in creating outreach interventions and informing risk stratification. The study also seeks to determine whether skin care knowledge varies by adherence to masculine norms. This knowledge can be used to guide patient education in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 or older
* Subjects identity as Male
* Reside in the United States
* Able to complete an online survey published in English

Exclusion Criteria:

- Subjects who do not meet the inclusion criteria - Subjects who have previously completed the study

Ages: 18 Years to 125 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult men residing in the United States
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Frequency of skin care behaviors | 2 months
  Research participants will be assigned masculinity classifications based on their Avoidance to femininity subscores. The frequency at which research participants in each masculinity class practice the skin care behaviors assessed in the questionnaire will be reported. The unit of measure will be a numerical value, number of participants.
Number of participants with certain skin care attitudes | 2 months
  Research participants will be assigned masculinity classifications based on their Avoidance to femininity subscores. The study will also report the number of participants in each masculinity class with specific skin care attitudes. The unit of measure will be a numerical value, number of participants.
Skin Care Knowledge Scores | 2 months
  Research participants will be assigned masculinity classifications based on their Avoidance to femininity subscores. Skin care knowledge scores for each masculinity class will also be reported. The unit of measure will be a numerical value, raw score.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Connell, R.W.Beth 1987. Gender and power. Sydney, Australia: Allen, Mercer and Urwin.
- [Background] David, D. S., & Brannon, R 1976. The Forty-nine percent majority: the male sex role. New York: Random House.
- [Background] Robertson, S. 2007. Understanding men and health: masculinities, identity, and well-being. Milton Keynes: Open University Press.
- [Background] Griffith, D. M., Gilbert, K. L., Bruce, M. A., & Thorpe, R. J. (2016). Masculinity in Men's Health: Barrier or Portal to Healthcare? Men's Health in Primary Care, 19-31.
- [Background] Levant RF, Hall RJ, Rankin TJ. Male Role Norms Inventory-Short Form (MRNI-SF): development, confirmatory factor analytic investigation of structure, and measurement invariance across gender. J Couns Psychol. 2013 Apr;60(2):228-238. doi: 10.1037/a0031545. Epub 2013 Feb 18. PMID 23421776
- [Background] Griffith DM, Gunter K, Watkins DC. Measuring masculinity in research on men of color: findings and future directions. Am J Public Health. 2012 May;102 Suppl 2(Suppl 2):S187-94. doi: 10.2105/AJPH.2012.300715. Epub 2012 Mar 8. PMID 22401519
- [Background] American Academy of Dermatology. Skin care tips for men. Retrieved March 04, 2017, from https://www.aad.org/public/skin-hair-nails/skin-care/skin-care-for-men
- [Background] American Academy of Dermatology. SPOTme Skin Cancer Quiz. Retrieved March 04, 2017, from https://www.aad.org/public/spot-skin-cancer/programs/screenings/spotme-skin-cancerquiz